CLINICAL TRIAL: NCT04718844
Title: A Randomised, Single-blind, Placebo-controlled, Phase 1, Single-ascending and Multiple-dose Study in Adult Subjects With Alpha/Beta-thalassaemia and Very Low- and Low-risk Myelodysplastic Syndrome to Investigate the Safety, Tolerability, Pharmacokinetic, and Pharmacodynamic Response of SLN124.
Brief Title: A Study Investigate the Safety, Tolerability, Pharmacokinetic, and Pharmacodynamic Response of SLN124 in Adults With Alpha/Beta-thalassaemia and Very Low- and Low-risk Myelodysplastic Syndrome
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Silence Therapeutics plc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SLN124-002
Record Dates: First submitted 2021-01-19; First posted 2021-01-22 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2024-01

CONDITIONS: Non-transfusion-dependent Thalassemia; Low Risk Myelodysplastic Syndrome; Very-Low Risk Myelodysplastic Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (18):
- 1.0mg/kg - Thalassaemia (Experimental)
  Interventions: Drug: SLN124
- 3.0mg/kg - Thalassaemia (Experimental)
  Interventions: Drug: SLN124
- 6.0mg/kg - Thalassaemia (Experimental)
  Interventions: Drug: SLN124
- Placebo - Thalassaemia (Placebo Comparator)
  Interventions: Drug: Placebo
- Xmg/kg - Thalassaemia (Experimental)
  Interventions: Drug: SLN124
- 1.0mg/kg - Myelodysplastic Syndrome (Experimental)
  Interventions: Drug: SLN124
- 3.0mg/kg - Myelodysplastic Syndrome (Experimental)
  Interventions: Drug: SLN124
- 10.0mg/kg - Myelodysplastic Syndrome (Experimental)
  Interventions: Drug: SLN124
- Xmg/kg - Myelodysplastic Syndrome (Experimental)
  Interventions: Drug: SLN124
- 3.0mg/kg - Thalassaemia multi dose (Experimental)
  Interventions: Drug: SLN124
- 10.0mg/kg - Thalassaemia multi dose (Experimental)
  Interventions: Drug: SLN124
- Xmg/kg - Thalassaemia multi dose (Experimental)
  Interventions: Drug: SLN124
- 3.0mg/kg - Myelodysplastic Syndrome multi dose (Experimental)
  Interventions: Drug: SLN124
- 10.0mg/kg - Myelodysplastic Syndrome multi dose (Experimental)
  Interventions: Drug: SLN124
- Xmg/kg - Myelodysplastic Syndrome multi dose (Experimental)
  Interventions: Drug: SLN124
- Placebo - Thalassaemia multi dose (Placebo Comparator)
  Interventions: Drug: Placebo
- Placebo - Myelodysplastic Syndrome (Placebo Comparator)
  Interventions: Drug: Placebo
- Placebo - Myelodysplastic Syndrome multi dose (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SLN124 — SLN124 for subcutaneous (s.c.) injection
  Arms: 1.0mg/kg - Myelodysplastic Syndrome; 1.0mg/kg - Thalassaemia; 10.0mg/kg - Myelodysplastic Syndrome; 10.0mg/kg - Myelodysplastic Syndrome multi dose; 10.0mg/kg - Thalassaemia multi dose; 3.0mg/kg - Myelodysplastic Syndrome; 3.0mg/kg - Myelodysplastic Syndrome multi dose; 3.0mg/kg - Thalassaemia; 3.0mg/kg - Thalassaemia multi dose; 6.0mg/kg - Thalassaemia; Xmg/kg - Myelodysplastic Syndrome; Xmg/kg - Myelodysplastic Syndrome multi dose; Xmg/kg - Thalassaemia; Xmg/kg - Thalassaemia multi dose
Drug: Placebo — Sodium chloride for s.c. injection
  Arms: Placebo - Myelodysplastic Syndrome; Placebo - Myelodysplastic Syndrome multi dose; Placebo - Thalassaemia; Placebo - Thalassaemia multi dose

SUMMARY:
This study will investigate the safety and tolerability of SLN124 in patients with Thalassaemia or patients with Very Low- and Low-risk Myelodysplastic Syndrome (MDS) after single ascending s.c. doses and multiple doses in healthy male and female subjects. Up to 7 cohorts of 56 patients with Thalassaemia and up to 7 cohorts of 56 patients with MDS will be enrolled. Each subject will receive single or multiple doses of SLN124 or placebo given by subcutaneous (s.c) injection.

ELIGIBILITY:
Inclusion Criteria:

* Adult with alpha- or beta-thalassaemia or compound heterozygous haemoglobin E/beta-thalassaemia or adult with very low- or low-risk MDS according to the 2016 revision to the World Health Organisation classification.
* All subjects must agree to adhere to appropriate contraception requirements.
* Subjects must provide written informed consent and be able to comply with all study requirements.
* Body mass index ≥18 kg/m2 and ≤35 kg/m2 at screening.
* At least one of: a) Mean ferritin >250 μg/L based on a minimum of 2 measurements ≥1 week apart within 20 days before the planned dosing day, in the absence of active significant infection; b) Mean TSAT >40% measured on a minimum of 2 occasions ≥1 week apart within 20 days before the planned dosing day; c) Liver iron >3 mg Fe/g dry weight, measured according to local procedures.
* Mean baseline haemoglobin concentration ≥5 g/dL and ≤11 g/dL, based on a minimum of 2 measurements ≥1 week apart, within 20 days before the planned dosing day.

Exclusion criteria

* Adult with haemoglobin S/alpha-thalassaemia or haemoglobin S/beta-thalassaemia or adult with secondary MDS, i.e., MDS that is known to have arisen because of chemical injury or treatment with chemotherapy and/or radiation for another disease.
* History of multiple drug allergies or history of allergic reaction to an oligonucleotide or GalNAc, or intolerance to s.c. injections.
* Known infection with HIV, or active infectious hepatitis A, B, or C virus.
* Any conditions which, in the opinion of the Investigator, would make the subject unsuitable for enrolment in the study or could interfere with the subject's participation in, or completion of the study.
* History or clinical evidence of alcohol or illegal drug misuse within 2 years before screening.
* Currently using ESA, or plan to use ESA at any point during the study.
* Require daily treatment with 1 or more non-steroidal anti-inflammatory drugs during the study period. Paracetamol will be permitted for use as an antipyretic and/or analgesic.
* Treatment, or change in treatment with prohibited medications as specified in the protocol
* Treatment with ICT where the subject has not been on a stable dose for at least 8 weeks before screening or it is planned to initiate ICT therapy during the study.
* Clinically significant cardiac disease
* Clinically significant pulmonary disease

For subjects with thalassaemia:

* Treatment, or change in treatment with prohibited medications as specified in the protocol
* currently and anticipated to receiving more than 5 units of RBCs during the 24 weeks to 6 weeks period before first dose of study drug.

For subjects with very low / low-risk MDS:

* Previous allogeneic or autologous stem cell transplantation.
* Currently or planned to receive treatment with a corticosteroid for MDS within 8 weeks before screening.
* Currently or planned to receive treatment with haematopoietic growth factors (e.g., eltrombopag, romiplostim) within 8 weeks before screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2021-04-14 (Actual); Primary Completion 2023-05-23 (Actual); Study Completion 2023-05-23 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events | Day 84
  safety and tolerability will be reported separately following single-dose administration.
Incidence of treatment-emergent adverse events | Day 140
  safety and tolerability will be reported separately following multi-dose administration.

SECONDARY OUTCOMES:
Pharmacokinetic: peak plasma concentration (Cmax) | Day 84 and Day 140
  Will be reported separately following single-dose and multiple-dose administration.
Pharmacokinetic: area under the plasma concentration (AUC) | Day 84 and Day 140
  Will be reported separately following single-dose and multiple-dose administration.
Pharmacokinetic: apparent total clearance from plasma after s.c injection (CL/F) | Day 84 and Day 140
  Will be reported separately following single-dose and multiple-dose administration.
Pharmacodynamic biomarkers: Change in TSAT after s.c injection. | Day 84 and Day 140
  safety and tolerability will be reported separately following single-dose and multiple-dose administration.
Pharmacodynamic biomarkers: Change in hepcidin after s.c injection. | Day 84 and Day 140
  safety and tolerability will be reported separately following single-dose and multiple-dose administration.
Pharmacodynamic biomarkers: Change in serum iron after s.c injection. | Day 84 and Day 140
  safety and tolerability will be reported separately following single-dose and multiple-dose administration.
Pharmacodynamic biomarkers: Change in haemoglobin after s.c injection. | Day 84 and Day 140
  safety and tolerability will be reported separately following single-dose and multiple-dose administration.

CONTACTS AND LOCATIONS:
Locations (20):
- Germany (2):
  - Universitaetsklinikum Duesseldorf, Düsseldorf
  - Universitat Leipzig, Leipzig
- Israel (4):
  - Rambam Health Care Campus, Haifa
  - Sheba Medical Center, Ramat Gan
  - Bar-Ilan University - Faculty of Medicine, Safed
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (2):
  - AUSL della Romagna - Ospedale di Ravenna, Ravenna
  - Azienda Unità Sanitaria Locale - IRCCS di Reggio Emilia, Reggio Emilia
- Jordan (3):
  - Jordan University Hospital, Amman
  - King Hussein Cancer Center, Amman
  - Irbid Speciality Hospital, Irbid
- Malaysia (2):
  - Sarawak General Hospital, Kampung Sarawak
  - Hospital Ampang, Kampung Selangor
- Thailand (4):
  - King Chulalongkorn Memorial Hospital, Bangkok
  - Mahidol University - Faculty of Medicine - Ramathibodi Hospital, Bangkok
  - Mahidol University - Siriraj Hospital, Bangkok
  - Faculty of Medicine, Chiang Mai University, Chiang Mai
- United Kingdom (3):
  - University Hospital of Wales, Cardiff
  - The Leeds Teaching Hospitals NHS Trust - Saint James's University Hospital, Leeds
  - Hammersmith Medicines Research Ltd (HMR), London